CLINICAL TRIAL: NCT04859452
Title: A Four-part, Single-center, Open-label, Phase I Clinical Study to Evaluate the Drug-Drug Pharmacokinetic Interaction Between DBPR108 at Steady-state and Metformin Hydrochloride/Glibenclamide/Valsartan/ Simvastatin in Healthy Subjects
Brief Title: A Study to Evaluate the DDI of DBPR108 With Metformin,Glibenclamide,Valsartan, or Simvastatin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA1118-CSP-010
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — DBPR108; Metformin; Glyburide; Valsartan; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The DDI of DBPR108 tablets and Metformin hydrochloride tablets (Experimental): Subjects will receive a single dose of metformin hydrochloride on Day 1, then take once-daily DBPR108 100 mg on Day 4 through Day 8 and a single dose of metformin hydrochloride on Day 8.
  Interventions: Drug: DBPR108 tablets; Drug: Metformin hydrochloride tablets
- The DDI of DBPR108 tablets and Glibenclamide tablets (Experimental): Subjects will receive a single dose of Glibenclamide on Day 1, then take once-daily DBPR108 100 mg on Day 4 through Day 8 and a single dose of Glibenclamide on Day 8.
  Interventions: Drug: DBPR108 tablets; Drug: Glibenclamide tablets
- The DDI of DBPR108 tablets and Valsartan Capsules (Experimental): Subjects will receive a single dose of Valsartan on Day 1, then take once-daily DBPR108 100 mg on Day 4 through Day 8 and a single dose of Valsartan on Day 8.
  Interventions: Drug: DBPR108 tablets; Drug: Valsartan Capsules
- The DDI of DBPR108 tablets and Simvastatin tablets (Experimental): Subjects will receive a single dose of Simvastatin on Day 1, then take once-daily DBPR108 100 mg on Day 4 through Day 8 and a single dose of Simvastatin on Day 8.
  Interventions: Drug: DBPR108 tablets; Drug: Simvastatin tablets

INTERVENTIONS:
Drug: DBPR108 tablets — Drug: DBPR108, tablet, oral
  Other Names: DBPR108
Drug: Metformin hydrochloride tablets — Drug: Metformin hydrochloride, tablet, oral
  Arms: The DDI of DBPR108 tablets and Metformin hydrochloride tablets
Drug: Glibenclamide tablets — Drug: Glibenclamide, tablet, oral
  Arms: The DDI of DBPR108 tablets and Glibenclamide tablets
Drug: Valsartan Capsules — Drug: Valsartan, capsule, oral
  Arms: The DDI of DBPR108 tablets and Valsartan Capsules
Drug: Simvastatin tablets — Drug: Simvastatin, tablet, oral
  Arms: The DDI of DBPR108 tablets and Simvastatin tablets

SUMMARY:
This is a four-part, single-center, open-label, single-sequence crossover phase I clinical study to characterize the Drug-Drug Interaction (DDI) potential of DBPR108 at steady-state with Metformin hydrochloride, Glibenclamide, Valsartan, or Simvastatin in Healthy Subjects. This study also aims to evaluate the safety and tolerability of DBPR108 in the presence of Metformin hydrochloride, Glibenclamide, Valsartan, or Simvastatin.

DETAILED DESCRIPTION:
DBPR108 is a potent dipeptidylpeptidase-4 inhibitor. This study will be run in four parts to characterize the Drug-Drug Interaction (DDI) potential of DBPR108 with the expected concomitant drugs (Metformin hydrochloride, Glibenclamide, Valsartan, Simvastatin) in Healthy Subjects. Each part of this study consists of a screening period (Day -14 to Day -1), a baseline period (Day -1), a treatment period (Day 1 to Day 9), and a follow-up visit on Day 15. Approximately 14 subjects will be enrolled in each part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign the informed consent form, understand the trial procedures, and be willing to comply with all trial procedures and restrictions；
* 18 years to 45 years (inclusive), male or female；
* Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Body mass index (BMI) : 18-30 kg/m2 (inclusive) (BMI= weight (kg)/height 2 (m2))；
* Subjects (including partners) are willing to use effective contraceptives from screening to the 6 months after the last dose administration；
* Be judged to be in good health by the investigator, based on the physical examination, vital sign examination, 12-lead electrocardiogram (ECG) examination and laboratory examination；

Exclusion Criteria:

* Subjects who have a history of allergic conditions (such as asthma, urticaria), or have a history of allergy to two or more drugs or food, or may be allergic to the test drug and the related compounds;
* Have a history of severe diseases, such as cardiovascular, respiratory, liver, gastrointestinal, endocrine, hematologic, mental/nervous systems diseases within 1 year prior to screening；
* Subjects who have previously undergone surgery that may affect drug absorption, distribution, metabolism, or excretion (e.g., subtotal gastrectomy), or who have a scheduled surgical plan during the study period;
* Use of any prescription drug, over-the-counter drug, or herbal medicine within 2 weeks prior to screening;
* Drug abuse, or positive urine drug screen at screening；
* Smoking more than 5 cigarettes per day within 3 months prior to screening；
* Average alcohol intake is more than 28g alcohol (male) or 14g (female) per week (14g ≈ 497mL beer, or 44mL spirits with low alcohol content, or 145mL wine) within the 3 months prior to screening, or taking any alcohol within 48 hours before dosing, or a positive ethanol breath test at screening；
* Consumption of grapefruit juice, Methylxanthine-rich food or beverage (such as coffee, tea, cola, chocolate, energy drinks) within 48 hours before the administration, or have strenuous exercise, or have other factors affecting drug absorption, distribution, metabolism, excretion, etc；
* Participation in another clinical trial within 3 months before screening；
* Blood donation (or blood loss) ≥400 mL, or receiving whole blood transfusions or erythrocyte suspension transfusions within 3 months prior to the screening；
* The patients who have undergone comprehensive inspection with any significant clinical significant in physical examination (vital signs, physical examination), routine laboratory examination (blood routine, blood biochemical examination, urine routine), chest X-ray (anteroposterior), abdominal B (liver, bile, pancreas, spleen and kidney) and other examinations, as judged by the investigator;
* Have a positive test result of hepatitis B surface antigen, hepatitis C antibody, anti-human immunodeficiency virus antibody or anti-Treponema pallidum specific antibody;
* A pregnant/lactating woman, or has a positive pregnancy test at screening or during the trial.；
* Not suitable for this study as judged by the investigator；

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic parameters of Metformin, Glibenclamide, Valsartan, Simvastatin, Simvastatin acid and DBPR108 | Day 1 to Day 9
  Peak Plasma Concentration (Cmax)
The pharmacokinetic parameters of Metformin, Glibenclamide, Valsartan, Simvastatin, Simvastatin acid and DBPR108 | Day 1 to Day 9
  Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
The pharmacokinetic parameters | Day 1 to Day 9
  The pharmacokinetic parameters (Metformin, Glibenclamide, Valsartan, Simvastatin, Simvastatin acid, DBPR108) : Tmax
The pharmacokinetic parameters | Day 1 to Day 9
  The pharmacokinetic parameters (Metformin, Glibenclamide, Valsartan, Simvastatin, Simvastatin acid, DBPR108) : t1/2
The pharmacokinetic parameters | Day 1 to Day 9
  The pharmacokinetic parameters (Metformin, Glibenclamide, Valsartan, Simvastatin, Simvastatin acid, DBPR108) : Vz/F
The pharmacokinetic parameters | Day 1 to Day 9
  The pharmacokinetic parameters (Metformin, Glibenclamide, Valsartan, Simvastatin, Simvastatin acid, DBPR108) : CL/F
The number of volunteers with adverse events as a measure of safety and tolerability | Day 1 to Day 15
  The number of volunteers with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, China